CLINICAL TRIAL: NCT05105438
Title: Comparing Oral Iron Supplementation Using Alternate-day Dosing to the Standard of Care Consecutive-day Dosing in Iron-depleted Women With or Without Mild Anemia
Brief Title: Alternate Day vs. Daily Iron Supplementation in Iron Depleted Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Jessica Rigutto, Dr., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPS_CH
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia
Keywords: iron supplementation; dosing regimen; iron sulfate; women of reproductive age
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blinded randomized controlled study: participants and investigators are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consecutive Day Dosing (Active Comparator): 100 mg iron as FeSO4 daily for 3 months, followed by matched placebo daily for 3 months.
  Interventions: Dietary Supplement: Consecutive Day Dosing
- Alternate Day Dosing (Experimental): 100 mg iron as FeSO4 and matched placebo on alternating days for 6 months.
  Interventions: Dietary Supplement: Alternate Day Dosing

INTERVENTIONS:
Dietary Supplement: Consecutive Day Dosing — 100 mg iron as FeSO4 daily for 3 months, followed by matched placebo daily for 3 months.
  Arms: Consecutive Day Dosing
Dietary Supplement: Alternate Day Dosing — 100 mg iron as FeSO4 and matched placebo on alternating days for 6 months.
  Arms: Alternate Day Dosing

SUMMARY:
Iron deficiency (ID) with or without anemia is a major public health problem worldwide, especially in women of reproductive age. Iron supplementation can be an effective strategy to prevent and treat ID and iron deficiency anemia (IDA). Recent studies suggests that giving oral iron every other day would be an optimized dosing regimen with maximized absorption and a lower incidence of gastrointestinal side effects compared to consecutive day dosing. Long-term trials in which participants and investigators are blinded to the dosing interval with iron status and gastrointestinal side effects as study outcomes are needed.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old,
* SF levels <25 μg/L,
* Hb levels ≥ 11 g/dL
* Normal Body Mass Index (18.5-25 kg/m2),
* In possession of a mobile phone on which the study app can be loaded,
* Signed informed consent,
* Not mandatory (only for subgroup analysis): having participated in a former stable iron isotope study in our laboratory between 1-5 y ago

Exclusion Criteria:

* Elevated CRP > 5 mg/L,
* Any metabolic, gastrointestinal, kidney or chronic disease (self-reported) affecting iron metabolism,
* Continuous/long-term use of medication, which may interfere with iron absorption, gut physiology and iron metabolism,
* Consumption of additional iron supplements over the study period,
* Consumption of iron supplements since screening,
* Difficulties with blood sampling,
* Known hypersensitivity or allergy to iron or placebo capsules in the given amount (ferrous sulfate, mannitol, silica)
* Pregnancy, breastfeeding
* Women who intend to become pregnant during the course of the study,
* Known or suspected non-compliance, drug or alcohol (more than 2 drinks/day) abuse,
* Smokers (> 1 cigarette per week),
* Participant is likely to be absent on one the study appointments,
* Inability to follow the procedures of the study, e.g. due to language problems, self-reported psychological disorders, etc. of the participant.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 150 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Serum Ferritin (SF) | Day 93
  in consecutive day group
Serum Ferritin (SF) | Day 186
  in alternate day group
Event rate of GI side effects | Day 90
  in consecutive day group
Event rate of GI side effects | Day 183
  in alternate day group

SECONDARY OUTCOMES:
Hemoglobin (Hb) | Day 0
Hemoglobin (Hb) | Day 46
Hemoglobin (Hb) | Day 90
Hemoglobin (Hb) | Day 139
Hemoglobin (Hb) | Day 183
Serum Ferritin (SF) | Day 0
Serum Ferritin (SF) | Day 46
Serum Ferritin (SF) | Day 93
Serum Ferritin (SF) | Day 139
Serum Ferritin (SF) | Day 186
Serum Transferrin Receptor (sTfR) | Day 0
Serum Transferrin Receptor (sTfR) | Day 46
Serum Transferrin Receptor (sTfR) | Day 93
Serum Transferrin Receptor (sTfR) | Day 139
Serum Transferrin Receptor (sTfR) | Day 186
Total iron binding capacity (TIBC) | Day 0
Total iron binding capacity (TIBC) | Day 93
Total iron binding capacity (TIBC) | Day 186
Serum Iron (SFe) | Day 0
Serum Iron (SFe) | Day 93
Serum Iron (SFe) | Day 186
C-Reactive Protein (CRP) | Day 0
C-Reactive Protein (CRP) | Day 46
C-Reactive Protein (CRP) | Day 93
C-Reactive Protein (CRP) | Day 139
C-Reactive Protein (CRP) | Day 186
Alpha-1-acid Glycoprotein (AGP) | Day 0
Alpha-1-acid Glycoprotein (AGP) | Day 46
Alpha-1-acid Glycoprotein (AGP) | Day 93
Alpha-1-acid Glycoprotein (AGP) | Day 139
Alpha-1-acid Glycoprotein (AGP) | Day 186
Intestinal Fatty Acid-binding Protein (I-FABP) | Day 0
Intestinal Fatty Acid-binding Protein (I-FABP) | Day 90
Intestinal Fatty Acid-binding Protein (I-FABP) | Day 183
Calprotectin | Day 0
Calprotectin | Day 90
Calprotectin | Day 183
Hepcidin | Day 0
Hepcidin | Day 46
Hepcidin | Day 90
Hepcidin | Day 139
Hepcidin | Day 183
Event rate of GI side effects | Day 90
Event rate of GI side effects | Day 183
Incidence of GI side effects | Day 90
Incidence of GI side effects | Day 183
Event proportion of GI side effects | Day 90
Event proportion of GI side effects | Day 183
Severity of GI side effects | Day 90
Severity of GI side effects | Day 183
Fecal blood losses | Day 0
Fecal blood losses | Day 90
Fecal blood losses | Day 183
Iron absorption from supplements | Day 90
Iron absorption from supplements | Day 183

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stoffel, Dr., Principal Investigator — Human Nutrition Laboratory, ETH Zuerich
Locations (1):
- ETH Zurich; Human Nutrition Laboratory; Institute of Food, Nutrition and Health, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Siebenthal HK, Gessler S, Vallelian F, Steinwendner J, Kuenzi UM, Moretti D, Zimmermann MB, Stoffel NU. Alternate day versus consecutive day oral iron supplementation in iron-depleted women: a randomized double-blind placebo-controlled study. EClinicalMedicine. 2023 Nov 3;65:102286. doi: 10.1016/j.eclinm.2023.102286. eCollection 2023 Nov. PMID 38021373